CLINICAL TRIAL: NCT02334865
Title: A Phase I Study of Safety, Tolerability and Immunological Effects of SVN53-67/M57-KLH in Patients With Multiple Myeloma Receiving Lenalidomide Maintenance Therapy
Brief Title: SVN53-67/M57-KLH Peptide Vaccine in Treating Patients With Newly Diagnosed Multiple Myeloma Receiving Lenalidomide Maintenance Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 247913; NCI-2014-02621 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 247913 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Partial Response of Multiple Myeloma or Plasma Cell Leukemia; Plasma Cell Myeloma
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma | interventions — incomplete Freund's adjuvant; montanide ISA 51; Lenalidomide; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (vaccine and week-4 lenalidomide maintenance therapy) (Experimental): Patients receive SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant SC and sargramostim SC every 2 weeks at weeks 0, 2, 4, and 6 for up to 4 doses and then receive a booster in week 12. Beginning in week 4, patients receive lenalidomide maintenance therapy PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Incomplete Freund's Adjuvant; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine
- Group B (vaccine and week-0 lenalidomide maintenance therapy) (Experimental): Patients receive SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant SC and sargramostim SC every 2 weeks at weeks 4, 6, 8, and 10 for up to 4 doses and then receive a booster in week 16. Beginning in week 0, patients receive lenalidomide maintenance therapy PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Incomplete Freund's Adjuvant; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Sargramostim; Biological: SVN53-67/M57-KLH Peptide Vaccine

INTERVENTIONS:
Biological: Incomplete Freund's Adjuvant — Given SC
  Other Names: Freund's Incomplete Adjuvant; IFA; ISA-51; Montanide ISA 51; Montanide ISA-51
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Biological: SVN53-67/M57-KLH Peptide Vaccine — Given SC

SUMMARY:
This phase I trial studies the safety of SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant together with sargramostim in treating patients with newly diagnosed multiple myeloma who are receiving lenalidomide maintenance therapy. Vaccines made from survivin peptide may help the body build an effective immune response to kill cancer cells that express survivin. Incomplete Freund's adjuvant may help stimulate the body's immune response to a vaccine treatment. Colony-stimulating factors, such as sargramostim, may increase the production of blood cells. Lenalidomide may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant and sargramostim before or after the start of lenalidomide maintenance therapy may be a better treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity profile of the SVN53-67/M57-KLH peptide (SVN53-67/M57-KLH peptide vaccine) in Montanide ISA 51 (incomplete Freund's adjuvant) plus GM-CSF (sargramostim) (vaccine), given before or after the start of lenalidomide maintenance in patients with multiple myeloma.

SECONDARY OBJECTIVES:

I. To measure the immune responses induced by SVN53-67/M57-KLH with Montanide ISA 51 plus GM-CSF, either alone or with lenalidomide maintenance added either before or after the vaccine.

TERTIARY OBJECTIVES:

I. To collect preliminary data on therapeutic efficacy of this combination against multiple myeloma, including response rate, time to progression and disease progression slope.

II. To test if human leukocyte antigen (HLA) types and survivin positivity affect the immune responses induced by SVN53-67/M57-KLH with Montanide ISA 51 plus GM-CSF.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant subcutaneously (SC) and sargramostim SC every 2 weeks at weeks 0, 2, 4, and 6 for up to 4 doses and then receive a booster in week 12. Beginning in week 4, patients receive lenalidomide maintenance therapy orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant SC and sargramostim SC every 2 weeks at weeks 4, 6, 8, and 10 for up to 4 doses and then receive a booster in week 16. Beginning in week 0, patients receive lenalidomide maintenance therapy PO QD in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 16, 20, and 24 weeks and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to adhere to the study visit schedule and other protocol requirements
* Patients with newly diagnosed multiple myeloma who have at least a partial response after induction therapy based on the International Working Group (IWG) Uniform Response Criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Must be free of systemic infection; subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection; subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment
* Absolute neutrophil count >= 750/mm^3
* Platelet count >= 30,000/mm^3
* Creatinine clearance >= 30 mL/minutes
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN)
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS)®, and be willing and able to comply with the requirements of the Revlimid REMS®
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program
* Able to take aspirin (81 or 325 mg) daily for prophylactic anticoagulation (patients intolerant to acetylsalicylic acid, ASA, may use warfarin or low molecular weight heparin or other anticoagulants as deemed appropriate by physician)
* Disease free of prior malignancies for > 2 years with exception of currently treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* All study participants must have one of the HLA alleles: HLA-A*02, HLA-A*03, HLAA*11, or HLA-A*24
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females; (lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study as determined by the Principal Investigator
* Chemotherapy, immunotherapy, radiotherapy, radiosurgery, interferon (e.g. Intron-A®), allergy desensitization injections, growth factors (e.g. Procrit®, Aranesp®, Neulasta®), interleukins (e.g. Proleukin®) or any investigational therapeutic medication within 4 weeks of study entry
* Known hypersensitivity to thalidomide, lenalidomide, Keyhole Limpet Hemocyanin (KLH), or granulocyte colony-macrophage stimulating factor (GM-CSF)
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive because of hepatitis B virus vaccine are eligible
* Any prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy or autoimmune disorders with visceral involvement
* Patients with a known diagnosis of plasma cell leukemia
* Systemic corticosteroid therapy > 2 mg of dexamethasone or equivalent per day at study entry
* Patients had prior autologous or allogeneic stem cell transplant; prior stem cell collection is allowed
* Life expectancy less than 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of the SVN53-67/M57-KLH peptide vaccine in incomplete Freund's adjuvant plus sargramostim, given before or after the start of lenalidomide maintenance | Up to 24 weeks
  The National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 will be used to evaluate toxicity. The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. The frequency of toxicities will also be tabulated for the regimen estimated to be the regimen-limiting toxicity.

SECONDARY OUTCOMES:
Immune response using interferon (IFN)-gamma enzyme-linked immunospot (ELISPOT) and multimer assays | Up to 24 weeks
  A responder is defined as a patient who has responded in either IFN-gamma ELISPOT or multimer assays. For both the ELISPOT and multimer assays, time course and magnitude of responses will be plotted and data will be treated using mixed-effect modeling. In addition, Kendall's tau-b will be used to determine whether ELISPOT and multimer responses are associated.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York